CLINICAL TRIAL: NCT07045623
Title: Comparison of Intensive Versus Standard Care & Education for Dyslipidemia in Hypertension and Diabetes Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Collaborators: Hanam City Center for Hypertension and Diabetes Registration (Unknown); Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VC25OISI0048
Record Dates: First submitted 2025-03-24; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Diabetes Mellitus; Dyslipidemia; Primary Prevention
Keywords: Primary prevention; Chronic disease; Dyslipidemia
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Dyslipidemias; Chronic Disease

STUDY DESIGN:
Intervention Model Description: A total of 348 participants will be enrolled, with 174 assigned to the intensive care and education group and 174 to the conventional care and education group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive Care and Education Group (Experimental): Through a visit to the center in 0 months, two instructors, one nurse and one nutritionist, provide an hour of diabetes and high blood pressure 1:15 group education, and an additional hour of lipid abnormalities and effects 1:15 group education. A total of two hours of education will be conducted, and the same content of lipid abnormality education conducted in 0 months will be conducted for an hour through visits in the third month. Hyperlipidemia education is conducted in the form of 1:15 small group education with the same content conducted in 0 months or 1:87 size group education. In particular, 1:87 form of large-scale education will be operated as a dialogue-oriented lecture that asks and answers questions, and will be conducted by doctors. In addition, in two months and four months, education on diabetes, high blood pressure, and dyslipidemia will be conducted briefly for three minutes through non-face-to-face management phone calls, not visits.
  Interventions: Other: centralized management and education group
- Standard Care and Education Group (No Intervention): For only 0 months, two instructors, one nurse and one nutritionist, will provide 1 hour of diabetes and high blood pressure 1:15 group education, which corresponds to standard management education.

INTERVENTIONS:
Other: centralized management and education group — If assigned to the test group (centralized management and education group), two instructors, one nurse and one nutritionist, will receive an hour of diabetes and high blood pressure 1:15, and will receive an hour of lipid disorder disease and impact 1:15 group education. You will receive a total of 2 hours of education, and you will receive 1 hour of lipid abnormality education conducted in 0 months through a visit in the third month. The dyslipidemia education was conducted in the form of 1:15 small group education or 1:87 group education, which was conducted in 0 months. In particular, the 1:87 form of large-scale education will be operated as a dialogue-oriented lecture that asks and answers questions, and will be conducted by doctors. And in 2 months and 4 months, education on diabetes, high blood pressure, and dyslipidemia will be shortened for 3 minutes through non-face-to-face management phone calls, not face-to-face.
  Arms: Intensive Care and Education Group

SUMMARY:
The prevalence of dyslipidemia is high among patients with hypertension and diabetes mellitus, which increases the risk of cardiovascular disease. However, many patients lack awareness and adherence to treatment and lifestyle modifications. Therefore, a more structured and intensive approach to management and education is required.

This study aims to implement intensive dyslipidemia management and education for patients registered at the Hanam City Hypertension and Diabetes Education Center and evaluate changes in blood lipid levels accordingly. Additionally, the study will analyze the impact of intensive education on patients' quality of life, health behaviors, and treatment adherence, ultimately contributing to the development of effective management strategies.

DETAILED DESCRIPTION:
1. Necessity of Dyslipidemia Management Education for Patients with Hypertension and Diabetes :

   The prevalence of dyslipidemia is high among patients with hypertension and diabetes mellitus, making it a major risk factor for cardiovascular diseases. Previous studies have demonstrated that intensive dyslipidemia management plays a crucial role in preventing cardiovascular events. However, the level of education and management provided in primary healthcare settings remains unstandardized, and there is a lack of research validating the effectiveness of structured intensive management programs.

   Enhancing education on dyslipidemia is not merely a therapeutic intervention but a preventive measure that can contribute to long-term health improvements in patients. Lifestyle modifications reinforced through intensive education serve as a complementary approach to pharmacological treatment, ultimately reducing healthcare costs and enabling the efficient allocation of medical resources. Therefore, this study aims to evaluate the effectiveness of intensive dyslipidemia management and education for patients with hypertension and diabetes, providing evidence-based treatment strategies.
2. Objectives and Expected Outcomes :

The primary objective of this study is to assess the impact of intensive dyslipidemia education on improving blood lipid profiles in patients with hypertension and diabetes. Through this evaluation, the study seeks to contribute to the establishment of a more structured and standardized dyslipidemia management model within the existing chronic disease management system in Korea.

Additionally, this study aims to analyze the cost-benefit effect of enhanced education and examine its influence on reducing healthcare expenditures and improving long-term patient health management. Notably, dyslipidemia education has high feasibility for implementation in primary healthcare institutions and public health centers without requiring additional infrastructure, making it a highly practical intervention.

Furthermore, standardizing educational content alone is expected to yield positive effects on patient management, serving as a critical reference for future public health policy development. The findings of this study are anticipated to contribute to the revision of national dyslipidemia management guidelines and policymaking while enhancing the effectiveness of chronic disease management initiatives led by health authorities.

ELIGIBILITY:
Inclusion Criteria:

* Patients registered in the Hanam City Hypertension and Diabetes Program
* Adults aged 30 to 80 years
* Individuals who have provided written informed consent to participate in the study

Exclusion Criteria:

* Chronic kidney disease stage 4 or higher (eGFR <30 mL/min/1.73m²)
* Patients with liver cirrhosis or severe liver disease
* Patients with a history of acute coronary syndrome within the past 6 months
* Pregnant or breastfeeding women • Individuals with psychiatric disorders that may affect study participation

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total cholesterol, Triglyceride, HDL-cholesterol, LDL-cholesterol levels at 6 months | at baseline (pre-intervention) and at 6 months (after the intervention)
  Change from Baseline in Total cholesterol, Triglyceride, HDL-cholesterol, LDL-cholesterol levels at 6 months

SECONDARY OUTCOMES:
Change from Baseline in systolic blood pressure, diastolic blood pressure at 6 months | at baseline (pre-intervention) and at 6 months (after the intervention)
  Change from Baseline in systolic blood pressure, diastolic blood pressure at 6 months
Change from Baseline in HbA1c level at 6 months | at baseline (pre-intervention) and at 6 months (after the intervention)
  Change from Baseline in HbA1c level at 6 months
Change from Baseline in Quality of Life assessed by SF-36 at 6 months | at baseline (pre-intervention) and at 6 months
  Change from Baseline in Quality of Life assessed by SF-36 at 6 months
Change from Baseline in structured questionnaire assessing lifestyle (Physical activity, Dietary habits, Alcohol consumption, Smoking status) | at baseline (pre-intervention) and at 6 months
  Physical activity : Ordinal categorical variable (Number of days in the past week the participant exercised for ≥30 minutes to promote health (e.g., walking, aerobic, yoga, cycling, swimming)) Dietary habits (1) : Binary categorical variable (In the past month, did you eat breakfast on average ≥5 times per week?) Dietary habits (2) : Binary categorical variable (In the past month, did you consume processed foods (e.g., bread, chips, instant noodles, mix coffee, soda, sugary beverages) ≥ once per week on average?) Alcohol consumption : Ordinal categorical variable (Do you currently drink alcohol? -> 1 = Frequently, 2 = Rarely, 3 = Never) Smoking status : Categorical variable (Do you currently smoke? -> 1 = Yes, 2 = No, 3 = Former smoker (Stopped))

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Korea, ST. Vincent's Hospital., Gyeonggi-do, Suwon-si, South Korea